CLINICAL TRIAL: NCT04957524
Title: Transvaginal Electrical Stimulation for the Treatment of OAB-dry
Brief Title: TEST-ON - Does iStim Reduce Urinary Urgency?
Acronym: TEST-ON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Anne Lenore Ackerman, Assistant Professor of Urology and Director of Research, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-005834
Record Dates: First submitted 2021-06-23; First posted 2021-07-12 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Overactive Bladder; Urgency-frequency Syndrome; Urinary Frequency More Than Once at Night
MeSH Terms: conditions — Urinary Bladder, Overactive; Nocturia

STUDY DESIGN:
Intervention Model Description: Patient will then be randomized to treatment A followed by treamtent B (Group 1) or treatment B followed by treatment A (Group 2).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be masked to which treatment they are receiving in which order. They will be randomly assigned to one of two groups. The randomization assignments will be generated by the principal statistician in the UCLA Department of Urology with a random number generator algorithm in Microsoft Excel so that the proposed recruited patients will be randomly assigned to control or intervention group in an equal amount per group. This will be stored in a central location on a password protected system on the UCLA Health Box for the research staff to access and as each patient is randomized they will use the next available group assignment on the sheet and cross them off. This will be closely monitored to maintain appropriate use. The randomization will occur at the time of enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Set Amplitude (Active Comparator): This arm is to test a specific amplitude. Participants will be instructed to set the amplitude to 20 mA, frequency to 20 Hz, and pulse duration to 5 mS. The parameters will stay the same for the entire session. This stimulation will last 15 minutes and patients will be instructed to perform the at-home therapy once per day.
  Interventions: Device: iStim TENS unit and Transvaginal Probe
- Customizable Amplitude (Experimental): In this arm, the participant will set the frequency to 12 Hz and pulse duration to 1 millisecond. The participant will be instructed to increase the amplitude gradually and set it at the maximal tolerable amplitude. This stimulation will last 15 minutes and patients will be instructed to perform the at-home therapy once per day.
  Interventions: Device: iStim TENS unit and Transvaginal Probe

INTERVENTIONS:
Device: iStim TENS unit and Transvaginal Probe — iStim TENS unit and Transvaginal Probe are both commercially available products. TENS units work by delivering small electrical impulses through electrodes either attached to the skin or through a transvaginal probe.
  iStim transvaginal probe will be inserted vaginally to provide transvaginal electrical stimulation.

SUMMARY:
Overactive bladder (OAB) is a chronic disorder with an overall prevalence in the adult population of over 10%, but that may exceed 40% in elderly groups. Most overactive bladder treatments are aimed at decreasing urgency incontinence episodes. The purpose of this study is to determine whether an at-home transvaginal electrical stimulation (TES) program works to alleviate symptoms of urgency in patients with urinary urgency and frequency without incontinence. This is a cross-over trial. Women >18 yo presenting with OAB-dry will be randomized to receive one of two TES at home programs for 4 weeks. After completion of the program, the participant's symptoms will be assessed with standardized patient questionnaires. There will then be a 3 week washout period followed by the second at-home TES program. At the completion of the second program, the participant's symptoms will be assessed with the same standardized questionnaires. The participants will be followed for 6 months following the completion of the TES program.

DETAILED DESCRIPTION:
This will be a prospective randomized cross over trial. We will recruit women who present to clinic to see a Female Pelvic Medicine and Reconstructive Surgery, fellowship-trained provider within the UCLA Health System with the symptoms of OAB-dry and have failed or decline anti-cholinergic therapy.

Screening: Patients will be made aware of the study by their physician. Interested subjects will interact with study staff in person or by telephone for a complete description of the study. If they wish to continue, they will be screened for eligibility by study staff. If eligible, they will be given as much time as they wish to complete the process of informed consent and have their questions answered. Consent will be obtained electronically using the RedCap system.

After informed consent, subjects will be asked to complete intake questionnaires, sent through the RedCap site. These questionnaires include the International Consultation on Incontinence Questionnaire-Female Lower Urinary Tract Symptoms (ICIQ-FLUTS), female GenitoUrinary Pain Index (fGUPI), Pelvic Organ Prolapse Distress Inventory (POPDI-6) portion of the Pelvic Floor Disability Index (PFDI), the first 8 questions of the OverActive Bladder questionnaire (OAB-q), the last question of the AUA symptom score, and the Urgency Perception Scale: UPC.

After informed consent, study staff will access subjects' medical records to obtain the results of standard care procedures that are regularly performed for patients with this symptomatology, specifically, pelvic exam and urodynamics.

Participants will be asked to make a research visit for training and to obtain materials. They will be issued the iStim device. Both groups will be oriented to the vaginal stimulation device which includes the iStim TENS unit and Transvaginal Probe. The iStim TENS unit delivers a bipolar square wave that can be delivered over a range of 0 to 100 mA. On the TENS unit the patient can set frequency, duration of stimulation, pulse duration, and amplitude. During each participant's in-person visit they will be instructed by trained study staff on how to use the electrical stimulation.

Patients will be randomized to treatment A followed by treatment B (Group 1) or treatment B followed by treatment A (Group 2). The patients will be blinded to which treatment they are receiving first.

Each treatment phase will be 4 weeks in duration. The washout period between phases will be three weeks. Patients will be given a log to record each session completed at home in order to determine compliance. They will also be asked to record the amplitude achieved for each session in the treatment phase. Patients will be able to report adverse events electronically through RedCap or by contacting study staff directly.

At the end of each 4-week treatment patients will be asked to complete the same intake questionnaires again with the addition of the select questions from the modified version of the Overactive Bladder Patient Satisfaction with Treatment Questionnaire (OAB-PSTQ) and Patient Global Assessment (PGA) which assesses their perception of the intervention.

At the end of the intervention, participants will be asked to complete a bladder diary again using the same IUGA bladder diary.

Participants will be followed through their medical record for 6 months after completion of study activities. Further OAB therapies tried will be recorded as well as pelvic exams and/or urodynamics done as part of their standard care. They will be asked to complete the set of intake questionnaires once more at the end of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age > 18 years old
* English speaking
* OAB symptoms for greater than 3 months duration defined as:
* Urgency: Answer to OAB-q3 > 4]
* Frequency: greater than 8 voids on bladder diary during waking hours and OAB-q1 > 3
* No urinary urge incontinence: OAB-q8 < 2 and OAB-q4 < 2
* No significant pelvic pain: fGUPI4 < 4

Exclusion Criteria:

* Age less than 18
* Pregnancy
* Vaginal infection or lesion
* Neurogenic bladder
* Immunocompromised state (hx of transplant, on immunosuppressing drugs)
* PVR >150cc
* Urinary tract infections
* Neurogenic bladder
* Reduced perception of vaginal sensation
* Metallic implants
* Implanted electrical devices (i.e. pace maker)

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Urinary urgency | This will be the difference in score from the date of enrollment to the end of both treatment arms. This will range from 11 weeks to 20 weeks.
  The primary outcome is the change in participant's reported urgency as measured by the composite score of the first 8 questions of the OAB-q questionnaire. The questionnaire is out of 8 with higher scores corresponding with more bother from urinary urgency. The primary outcome is the difference between the pre-treament and post-treatment scores. The range is 0 to 48 with a larger difference corresponding to more improvement in patient's urgency over the study period.

SECONDARY OUTCOMES:
Percentage of assigned treatment sessions that were successfully completed | 4 weeks
  Number of home programs completed compared to planned treatments based on paper treatment log completed by patient. Range is 0 to 100% completion.
Change in Urinary Urgency Episodes | This will be the difference in score from the date of enrollment to the end of both treatment arms. This will range from 11 weeks to 20 weeks.
  Change in number of urgency episodes (per 24 hours) as measured on the voiding diaries. This will be the difference in number of urgency episodes pretreatment compared to posttreatment. The range is 0 to 10 urgency episodes.
Change in number of micturitions per 24 hours | This will be the difference in score from the date of enrollment to the end of both treatment arms. This will range from 11 weeks to 20 weeks.
  Change in number of micturition episodes (per 24 hours) as measured on the voiding diaries. This will be the difference in number of micturition episodes pretreatment compared to post-treatment. The range is 0 to 20 micturition episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Anne L Ackerman, MD, PhD, Principal Investigator — UCLA, Department of Urology
Locations (1):
- UCLA Center for Women's Pelvic Health, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Yamanishi T, Yasuda K, Sakakibara R, Hattori T, Suda S. Randomized, double-blind study of electrical stimulation for urinary incontinence due to detrusor overactivity. Urology. 2000 Mar;55(3):353-7. doi: 10.1016/s0090-4295(99)00476-8. PMID 10699609
- [Background] Soomro NA, Khadra MH, Robson W, Neal DE. A crossover randomized trial of transcutaneous electrical nerve stimulation and oxybutynin in patients with detrusor instability. J Urol. 2001 Jul;166(1):146-9. PMID 11435843
- [Background] Primus G, Kramer G. Maximal external electrical stimulation for treatment of neurogenic or non-neurogenic urgency and/or urge incontinence. Neurourol Urodyn. 1996;15(3):187-94. doi: 10.1002/(SICI)1520-6777(1996)15:33.0.CO;2-B. PMID 8732985
- [Background] Messelink EJ. The overactive bladder and the role of the pelvic floor muscles. BJU Int. 1999 Mar;83 Suppl 2:31-5. doi: 10.1046/j.1464-410x.83.s2.7.x. No abstract available. PMID 10210602
- [Background] Hoffman D. Understanding multisymptom presentations in chronic pelvic pain: the inter-relationships between the viscera and myofascial pelvic floor dysfunction. Curr Pain Headache Rep. 2011 Oct;15(5):343-6. doi: 10.1007/s11916-011-0215-1. PMID 21739128
- [Background] Guralnick ML, Kelly H, Engelke H, Koduri S, O'Connor RC. InTone: a novel pelvic floor rehabilitation device for urinary incontinence. Int Urogynecol J. 2015 Jan;26(1):99-106. doi: 10.1007/s00192-014-2476-9. Epub 2014 Jul 30. PMID 25074260
- [Background] Brubaker L, Benson JT, Bent A, Clark A, Shott S. Transvaginal electrical stimulation for female urinary incontinence. Am J Obstet Gynecol. 1997 Sep;177(3):536-40. doi: 10.1016/s0002-9378(97)70142-x. PMID 9322620
- [Background] Amaro JL, Gameiro MO, Kawano PR, Padovani CR. Intravaginal electrical stimulation: a randomized, double-blind study on the treatment of mixed urinary incontinence. Acta Obstet Gynecol Scand. 2006;85(5):619-22. doi: 10.1080/00016340500495058. PMID 16752244
- [Derived] Torosis M, Stothers L, Cisneros C, Dominique G, Lenore Ackerman A. Transvaginal Electrical Stimulation for Treatment of Overactive Bladder Without Incontinence: A Pilot Cross-Over Clinical Trial. Neurourol Urodyn. 2025 Jun;44(5):977-986. doi: 10.1002/nau.70034. Epub 2025 Mar 26. PMID 40135809